CLINICAL TRIAL: NCT05090215
Title: A Randomised Controlled Trial to Assess the Efficacy of a Postoperative Supervised Exercise Programme in Patients Who Have Undergone Elective Curative Surgery for Colorectal Cancer.
Brief Title: Supervised Exercise for Post-surgery Colorectal Cancer Patients
Acronym: POSTEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21058
Record Dates: First submitted 2021-09-28; First posted 2021-10-22 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms
Keywords: exercise; rehabilitation; postoperative; colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity | interventions — Resistance Training; Blood Specimen Collection; Exercise Test

STUDY DESIGN:
Intervention Model Description: Single centre randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: Randomization will occur using www.sealedenvelope.com. This will be performed by a member of the research team on the patient's first visit. Patients will not be blinded due to the active nature of the intervention. Any independent review performed of data will be done by a researcher who has been blinded to group allocation.
  All possible analysis will be done in a single blinded manner (e.g., analysis of ultrasound scans, CPET, blood samples etc).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention group (Active Comparator): 2 resistance training session per week using a home-based resistance training pack and 75 minutes of vigorous or 150 minutes of moderate aerobic exercise per week (as per UK government guidelines) for 12 weeks. They will have 4 assessment points, pre-op, prior to the start of the exercise programme postoperatively, at 6 weeks post commencement of exercise and at 12 weeks to conclude the study. The assessment will include bloods, cardiopulmonary exercise testing, muscle ultrasound to ascertain muscle structure, functional composite scores and quality of life questionnaires.
  Interventions: Behavioral: Aerobic and resistance training 12 week exercise programme; Diagnostic Test: Venous blood sampling; Diagnostic Test: Muscle Ultrasound; Diagnostic Test: Cardiopulmonary exercise testing (CPET); Behavioral: Quality of life questionnaire completion
- Control group (Placebo Comparator): This group will receive standard postoperative care. They will also have 4 assessment points, pre-op, prior to the start of their standard postoperative care, 6 and finally 12 weeks later to conclude the study. The assessment will include bloods, cardiopulmonary exercise testing, muscle ultrasound to ascertain muscle structure, functional composite scores and quality of life questionnaires.
  Interventions: Diagnostic Test: Venous blood sampling; Diagnostic Test: Muscle Ultrasound; Diagnostic Test: Cardiopulmonary exercise testing (CPET); Behavioral: Quality of life questionnaire completion

INTERVENTIONS:
Behavioral: Aerobic and resistance training 12 week exercise programme — See arm/group description
  Arms: Exercise intervention group
Diagnostic Test: Venous blood sampling — full blood count, urea & electrolytes, C-reactive protein, coagulation screen, liver function tests, erythrocyte sedimentation rate.
Diagnostic Test: Muscle Ultrasound — Ultrasound of vastus lateralis to ascertain muscle structure (thickness, pennation angle and fascicle length)
Diagnostic Test: Cardiopulmonary exercise testing (CPET) — The assessment of anaerobic threshold as a measure of changes in aerobic function between the two groups will be assessed using CPET
Behavioral: Quality of life questionnaire completion — The use of validated questionnaires to assess quality of life parameters; Duke Activity Status Index (DASI), EORTC-QLQ C30 (quality of life for cancer patients) and the International Physical Activity Questionnaire (IPAQ).

SUMMARY:
Participants will undergo preoperative baseline screening and will be randomised to either normal postoperative care or a 12-week supervised exercise programme comprising of both an aerobic and resistance component

They will be assessed prior to surgery which will include cardiopulmonary exercise testing (CPET). This is a well-established method of assessing aerobic exercise response and is widely used in the perioperative period for assessment of cancer patients with co-morbidity. The assessment days will also include:

* muscle ultrasound (vastus lateralis) to ascertain muscle structure (thickness, pennation angle and fascicle length),
* blood tests,
* functional composite scores,
* quality of life questionnaires,

The assessment days will be carried out at four time points during the study; prior to surgery, before commencement of the exercise program, halfway through the intervention (6 weeks post commencement of exercise) and at the end of the study. In the week before the assessment days patients will wear a physical activity monitor to characterise their daily movements. The control group will also be assessed at the same time points and wear the activity monitors but will not take part in the exercise program.

All participants will have a physical activity monitor placed onto the right thigh in the midline at postoperative day 1 until discharge or day 7, whichever is sooner. This is a non-invasive measure of activity and can discriminate between whether a patient is lying, sitting, standing or walking.

Once participants self-report feeling able to start exercising again post-discharge, they will commence the 12 week programme. The intervention will consist of 2 resistance training (RET) sessions per week and 75 minutes of vigorous or 150 minutes of moderate aerobic exercise per week (can be split according to patient preference). They will receive a diary to log their sessions and will be monitored via twice weekly virtual follow-up (either telephone or video calling) and for the first 6 weeks weekly visits to ensure that they are adherent to the exercise protocol and provide any support/advice. Satisfactory compliance with the programme will be considered to be the completion of at least 27 sessions over the 12 week period, with a minimum of 13 out of 18 and 14 out of 18 sessions completed in the first and last 6 weeks, respectively.

DETAILED DESCRIPTION:
The study aims to provide a structured exercise programme to investigate whether a structured exercise programme following discharge from hospital will aid return to full activity. Exercise programmes are a well-tested and effective method of improving fitness in the healthy population. The government guidelines for adults aged 19 and above are to do at least 150 minutes of moderate intensity or 75 minutes of vigorous activity a week which can be split over multiple days. This does not require specialist equipment or costly interventions and include simple measures such as brisk walks and lifting weights. In conjunction with set resistance exercises, the investigators aim to use this as the target to provide a regimen that reaches this target for patients. Physical activity will also be measured at four timepoints during the study using a non-invasive physical activity monitor (ActivPAL) to compare between the intervention and control group.

Recruitment Understandably for the potential recruits this will be a difficult and emotional time period given their significant diagnosis that will have been given very soon prior to the research team's first interaction with them. Participants will be recruited in the outpatient setting but after the diagnosis and treatment plan has been made and conveyed by their parent team. Patients will be given all the information and at least 48 hours to consider their involvement in the study. They will then be re-contacted them via telephone and if they agree, researchers who are trained in taking consent will complete the consent process with the patient. No patients will be included who lack capacity or are in any other way unable to give informed consent. The research group have previously recruited for several prehabilitation studies in this way with good patient feedback and no reports of psychological harm.

Exercise

These guidelines are suitable for older participants with necessary adaptations. However, it is assumed that a small number older of participants may struggle to achieve these targets as they were not achievable for them prior to diagnosis and surgery. The investigators have a long and safe track record of exercise in the elderly in studies performed by the group, and clinical researchers will closely supervise the CPET. Unfamiliarity with exercise in itself is not a reason for non-inclusion in the study, but a more graduated increase in effort may be required for individual participants. There are clear inclusion and exclusion criteria outlined to minimise the risk of adverse outcomes following exercise in the participants. Cardiopulmonary exercise testing (CPET) will be included in the functional assessments at four points during the study. There is a theoretical risk of exercise-induced pathology that may occur secondary to this. The guidelines will be followed for absolute contraindications as laid out by the POETTS consensus guidelines (2018) and ATS/ACCP statement on CPET (2003). These include but are not limited to:

* Acute myocardial infarction (3-5 days)
* Unstable angina
* Uncontrolled arrhythmias causing symptoms or hemodynamic compromise (200 mm Hg systolic, 120 mm Hg diastolic)
* Syncope
* Active endocarditis
* Acute myocarditis or pericarditis
* Symptomatic severe aortic stenosis
* Uncontrolled heart failure
* Acute pulmonary embolus or pulmonary infarction
* Thrombosis of lower extremities
* Suspected dissecting aneurysm
* Uncontrolled asthma
* Pulmonary edema
* Room air desaturation at rest
* Respiratory failure
* Acute non cardiopulmonary disorder that may affect exercise performance or be aggravated by exercise (i.e. infection, renal failure, thyrotoxicosis)
* Mental impairment leading to inability to cooperate These patients will not be included in the study. Also, any abnormal results picked up at screening will warrant exclusion from the study, and the PI will communicate these to the participants' GP.

If any of the following occur both during exercise or CPET testing the programme will be terminated immediately and the participant withdrawn:

* Chest pain suggestive of ischaemia
* Ischemic ECG changes
* Complex ectopy
* Second or third degree heart block
* Fall in systolic pressure 20 mm Hg from the highest value during the test
* Hypertension (250 mm Hg systolic; 120 mm Hg diastolic)
* Severe desaturation: SpO2 ≤ 80% when accompanied by symptoms and signs of severe hypoxemia
* Sudden pallor
* Loss of coordination
* Mental confusion
* Dizziness or faintness
* Signs of respiratory failure CPET testing is the standard test for qualification of lack of cardiorespiratory fitness before operation and is used to stratify risk in higher risk patients as standard of care in the UK.

These guidelines will also be applied to those performing alternative forms of exercise such as brisk walking/running and resistance exercises. The resistance exercise component will via the use of resistance bands and therefore does not require equipment such as weight machines or free weights which can cause injury if applied incorrectly.

Those who volunteer for the study may be more active by virtue of a desire to be included. There is the potential for outcomes not being as generalizable to the whole population regardless of pre-existing physical activity, and also, impact of interventions may be lessened as both groups may be more fit than some groups of those who present for surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over MDT outcome of proven or high clinical suspicion of colorectal cancer Due to undergo either laparoscopic, robotic or open resection with curative intent Ability to exercise on a static bike (in order to complete the CPET, not required for the exercise programme) Ability to give informed consent Must be able to their organize own transport to RDH for the duration of the study in order to complete the supervised exercise sessions Availability for the period of study inclusion

Exclusion Criteria:

* Participants who lack capacity to consent Participants with a new diagnosis undergoing emergency surgery

Participants with a past medical history including the following:

* Recent myocardial infarction (MI) in the last 6 months or unstable angina Heart failure (New York Heart Association Class III/IV)
* Uncontrolled hypertension (BP>160/100)
* Previous stroke/TIA
* Cerebral or abdominal aortic aneurysm
* Severe respiratory disease including known pulmonary hypertension (>25mmHg)
* Exercise induced asthma or brittle asthma Abnormal blood and/or ECG results Patients who are unable to undergo CPET according to the Perioperative Exercise Testing and Training Society (POETTS) published consensus guidelines on performing CPET

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2024-01-27 (Actual); Study Completion 2024-01-27 (Actual)

PRIMARY OUTCOMES:
Anaerobic threshold change | 12 weeks from the commencement of the exercise programme
  To achieve a significant increase in anaerobic threshold (AT) on CPET (above 2.26ml/kg/min) in a cohort of colorectal cancer patients who have undergone surgery with curative intent following a 12-week combined aerobic and resistance exercise program compared to control.

SECONDARY OUTCOMES:
To assess whether all participants are able to complete the 12 week postoperative exercise programme (measured via study adherence and compliance) | 12 weeks from the commencement of the exercise programme
  To assess the feasibility of a twelve-week period of supervised exercise with a home-based component in this cohort of patients after surgery for colorectal cancer.
Quality of life improvements as reported by participants via validated questionnaires after application of a 12 week postoperative exercise programme | 12 weeks from the commencement of the exercise programme
  To assess whether patients feel any emotional/qualitative benefit from a period of supervised exercise in order to help them return to their normal activities of daily living more quickly/at all. The questionnaires employed will be the DASI, EORTC QLQ C30 and IPAQ.
Measure any changes see to vastus lateralis muscle composition via ultrasound after application of a 12 week postoperative exercise programme | 12 weeks from the commencement of the exercise programme
  Using muscle ultrasound, measure any changes seen during the study with the application of a supervised postoperative exercise program compared to control (normal postoperative care).
Change to the values inflammatory markers using venous blood samples after the application of a 12 week postoperative exercise programme | 12 weeks from the commencement of the exercise programme
  Capture any changes seen during the study via venepuncture in the inflammatory markers with the application of a supervised postoperative exercise program compared to control (normal postoperative care).

CONTACTS AND LOCATIONS:
Overall Officials: Jon Lund, MD, FRCS, Principal Investigator — jon.lund@nottingham.ac.uk
Locations (1):
- University of Nottingham, Royal Derby Hospital, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blackwell JEM, Doleman B, Boereboom CL, Morton A, Williams S, Atherton P, Smith K, Williams JP, Phillips BE, Lund JN. High-intensity interval training produces a significant improvement in fitness in less than 31 days before surgery for urological cancer: a randomised control trial. Prostate Cancer Prostatic Dis. 2020 Dec;23(4):696-704. doi: 10.1038/s41391-020-0219-1. Epub 2020 Mar 10. PMID 32157250
- [Background] Levett DZH, Jack S, Swart M, Carlisle J, Wilson J, Snowden C, Riley M, Danjoux G, Ward SA, Older P, Grocott MPW; Perioperative Exercise Testing and Training Society (POETTS). Perioperative cardiopulmonary exercise testing (CPET): consensus clinical guidelines on indications, organization, conduct, and physiological interpretation. Br J Anaesth. 2018 Mar;120(3):484-500. doi: 10.1016/j.bja.2017.10.020. Epub 2017 Nov 24. PMID 29452805